CLINICAL TRIAL: NCT06801379
Title: A Novel Inhaled Formulation of Melatonin to Treat Adults With Insomnia Disorder: a Randomised Open-Label Crossover Trial
Brief Title: A Novel Inhaled Formulation of Melatonin to Treat Adults With Insomnia: Pharmacokinetic Study
Acronym: Mela-Nia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Woolcock Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Hui Xin Ong, Chief Scientific Officer, Principal Investigator, Senior Research Fellow, Woolcock Institute of Medical Research
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 520241811859849
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-07

CONDITIONS: Insomnia
Keywords: Melatonin; Insomnia; Pharmacokinetics; Inhaled Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: Randomised, open-label, crossover trial
Masking Description: As this trial is open-label, all study staff and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Melatonin Arm (Experimental): 100 µg daily of inhaled melatonin delivered by pressurized metered dose inhaler for two weeks before habitual bedtime.
  Interventions: Drug: Inhaled Melatonin (100 μg)
- Oral Melatonin Arm (Active Comparator): 4 mg daily of orally delivered melatonin tablets for two weeks before habitual bedtime.
  Interventions: Drug: Oral Melatonin (4 mg)

INTERVENTIONS:
Drug: Inhaled Melatonin (100 μg) — An orally inhaled formulation of melatonin delivered by pressurised metered dose inhaler (pMDI) to be taken before bedtime. The pMDI will deliver a total of 100 μg of inhaled melatonin (2 x 50 μg/actuation). The investigational product is produced under Good Manufacturing Practice by Ab Initio Pharma Pty Ltd, a GMP certified manufacturer of pharmaceutical products.
  Other Names: Melatonin; N-Acetyl-5-methoxytryptamine
  Arms: Inhaled Melatonin Arm
Drug: Oral Melatonin (4 mg) — Two orally ingested tablets each containing 2 mg of melatonin (4 mg total) to be taken before bedtime. The investigational product is manufactured under Good Manufacturing Practice and is compliant with the TGA Therapeutic Order #101 that stipulates quality control requirements for capsule and pill-based products used in Australia.
  Other Names: N-Acetyl-5-methoxytryptamine; Circadin; Melatonin
  Arms: Oral Melatonin Arm

SUMMARY:
The goal of this clinical trial is to explore the potential benefits of an inhaled version of melatonin compared to oral melatonin tablets on adults with insomnia. The main question the trial aims to answer: is the time required for inhaled melatonin to reach peak concentration in the blood and then be eliminated from body different to that of oral melatonin tablets, in adults with insomnia?

5 participants will:

* Visit the research institute for a screening visit and for a daytime visit to take a melatonin treatment then provide blood samples over the course of 8 hours for each study drug treatment (3 visits in total)
* Take 100 μg of inhaled melatonin (2 inhaler puffs) once
* Take a 4 mg of oral melatonin (2 tablets) once

DETAILED DESCRIPTION:
This is a randomised open-label cross-over study of an inhaled formulation of melatonin (100 µg) versus oral melatonin tablets (4 mg) in adults with insomnia. The experiments performed for this trial will examine the effects of inhaled and oral drug delivery on the uptake and clearance of inhaled and oral melatonin.

To be enrolled in the trial, participants are required to complete an online pre-screening survey. Eligible participants will be directed to a separate webpage where they will be invited to review and download the Participant Information Sheet (PIS) and asked to provide their contact details and consent for a follow up call/email from the research team to book in a screening visit. At the screening visit, the study team will explain the study to each participant and provide the opportunity to ask any questions. The study team will also ensure participants have had ample time prior to the visit to read and understand the PIS. The consent form will be signed by both the participant and a medical officer and participants. Once participants have joined the efficacy study, they will be randomised into their first treatment group; inhaled melatonin (100 µg) or oral melatonin tablets (4 mg).

Participants will attend the laboratory for a daytime visit where they take the treatment once in the morning then remain at the laboratory over an approximately 8-hour period, providing blood samples every fifteen minutes during the first hour then hourly until 8 hours have passed since treatment. Participants will also be asked to rate their sleepiness on the Karolinska Sleepiness Scale each time blood is collected. There will be a 1 week washout period between treatments.

The study will recruit primarily through social media advertisements. The study will be coordinated from the Woolcock Institute of Medical Research, Sydney, Macquarie University, NSW, 2113, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of insomnia disorder as defined by the DSM-5 (difficulty initiating or maintaining sleep or waking up too early for at least 3 nights per week, for at least 3 months, with adequate opportunity and circumstances for sleep and at least one daytime impairment related to the sleep difficulty) and a score ≥15 on the ISI.
* History of subjective sleep onset latency (sSOL) ≥30 minutes on at least 3 nights per week in the previous 4 weeks.
* Able to provide informed electronic consent.
* Fluent English literacy.
* Adults aged 55+ years old.

Exclusion Criteria:

* People highly dependent on medical care as determined by a medical officer.
* Untreated moderate-severe sleep apnoea as diagnosed using in-home wrist oximetry (oxygen desaturation index>15, ongoing effectively treated sleep apnoea with insomnia will be allowed).
* Circadian disorders, narcolepsy, severe restless legs syndrome, and REM sleep behaviour disorder or uncontrolled psychiatric disorders.
* History of attempted suicide or current suicide ideation (indicated by a score >0 on Q9 of the Patient Health Questionnaire-9) at pre-screening.
* Objective cognitive decline measured by scoring ≤26 on the Montreal Cognitive Assessment (MoCA)
* Regular shift work, jet lag or trans-meridian travel (over 2h time difference) in the past week before randomisation.
* Pregnancy or lactation. Female participants of childbearing potential with a fertile sexual partner must have a negative serum pregnancy test result at the screening visit. Women will be advised to use contraception for the duration of the study.
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical trial due to safety concerns or compliance with clinical study procedures.
* Currently participating in or has participated in a research study of an investigational agent or device within 4 weeks of enrolment.
* Ongoing use of anti-psychotic medication, bosentan, efavirenz, etravirine, modafinil, rifampin, carbamazepine or illicit stimulants.
* Regular use of hypnotics (including melatonin, valerian, kava, benzodiazepines and Z-drugs), and other medications that can cause additive sedation (e.g. sedating antihistamines, tricyclic antidepressants, antipsychotics) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Regular use of psychostimulants (e.g., dexamfetamine, lisdexamfetamine, methylphenidate) or non-amphetamine psychostimulants (e.g., armodafinil, modafinil, atomoxetine) within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Use of antidepressant medications for treatment of low mood for less than one year or dose changes (escalation or tapering) or change in antidepressant medications within the past year.
* Regular use opioids within 14 days or 4-5 half-lives (whichever is longer) of starting the clinical trial.
* Ongoing use of THC- or CBD-containing products within 14 days prior to the start of the trial.
* Dependence or any other drug or alcohol dependence within the past two years (alcohol to be limited to no more than 2 standard drinks per day during trial period).
* Regular use of drugs that are CYP1A2 inhibitors (e.g. amiodarone, cimetidine, ciprofloxacin, fluvoxamine) or CYP1A2 inducers (e.g. carbamazepine, phenobarbital, rifampin, tobacco).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time to maximum Melatonin concentration | 0-8 hours post-treatment.
  Time to peak concentration (Tmax) of blood-based melatonin, analysed by melatonin ELISA.

SECONDARY OUTCOMES:
Melatonin area under the curve | 0-8 hours post-treatment.
  Area under the curve (AUC) of blood-based melatonin analysed by melatonin ELISA.
Maximum blood-based melatonin concentration | 0-8 hours post-treatment.
  Maximum concentration (Cmax) of blood-based melatonin, analysed by melatonin ELISA.
Melatonin half-life | 0-8 hours post-treatment.
  Half-life (T½) of blood based melatonin, analysed by melatonin ELISA.
Daytime sleepiness | Collected at t0 then every fifteen minutes during the first hour post-treatment, then once hourly until 8 hours post-treatment.
  Participant subjective daytime sleepiness, determined by the Karolinska Sleepiness Scale, a 9-point Likert scale (ranging from "Extremely alert" = 1 to "Very sleepy, great effort to keep awake, fighting sleep" = 9).

CONTACTS AND LOCATIONS:
Overall Officials: Hui Xin Ong, PhD, Principal Investigator — Woolcock Institute of Medical Research; Ron Grunstein, MBBS MD PhD FRACP, Principal Investigator — Woolcock Institute of Medical Research
Locations (1):
- Woolcock Institute of Medical Research, Macquarie Park, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon reasonable request to the Principal Investigators.
Time Frame: Non-identifiable IPD will become available one year after the Actual Study Completion Date and will remain available for fifteen years.
Access Criteria: Following Macquarie University access terms, access restrictions will be limited to appropriate permission, project proposal and approved from the investigator team and data custodian. Any Recipients of the data must obtain project and HREC approval prior to mediated access. The Coordinating Principal Investigator, Dr. Hui Xin Ong, will be retain access the de-identified data, stored on the Macquarie University Research Data Repository (RDR).
URL: https://libguides.mq.edu.au/research_data_repository